CLINICAL TRIAL: NCT03150693
Title: A Phase III Trial to Evaluate the Efficacy of the Addition of Inotuzumab Ozogamicin (a Conjugated Anti-CD22 Monoclonal Antibody) to Frontline Therapy in Young Adults (Ages 18-39 Years) With Newly Diagnosed Precursor B-Cell ALL
Brief Title: Inotuzumab Ozogamicin and Frontline Chemotherapy in Treating Young Adults With Newly Diagnosed B Acute Lymphoblastic Leukemia
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Unacceptable Toxicity
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A041501; NCI-2016-01981 (Registry Identifier: Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Allopurinol; Cytarabine; Daunorubicin; Vincristine; Dexamethasone; pegaspargase; Methotrexate; Biopsy; Cyclophosphamide; Mercaptopurine; Rituximab; Doxorubicin; Thioguanine; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (frontline chemotherapy) (Active Comparator): See detailed description.
  Interventions: Drug: Allopurinol; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Vincristine Sulfate; Drug: Dexamethasone; Drug: Pegylated L-Asparaginase; Drug: Methotrexate; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Mercaptopurine; Biological: Rituximab; Drug: Thioguanine; Other: Laboratory Biomarker Analysis
- Arm II (frontline chemotherapy, inotuzumab ozogamicin) (Experimental): Patients receive inotuzumab ozogamicin IV on days 1, 8, and 15 and undergo bone marrow aspirate and biopsy on day 28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive remission consolidated chemotherapy, interim maintenance chemotherapy, delayed intensification, and maintenance therapy as in Arm I.
  Interventions: Drug: Allopurinol; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Vincristine Sulfate; Drug: Dexamethasone; Drug: Pegylated L-Asparaginase; Drug: Methotrexate; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Mercaptopurine; Biological: Rituximab; Drug: Doxorubicin; Drug: Thioguanine; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Allopurinol — Given PO
Drug: Cytarabine — Given IT, IV, SC
Drug: Daunorubicin Hydrochloride — Given IV
Drug: Vincristine Sulfate — Given IV
Drug: Dexamethasone — Given PO or IV
Drug: Pegylated L-Asparaginase — Given IV
Drug: Methotrexate — Given IT, IV, PO
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cyclophosphamide — Given IV
Drug: Mercaptopurine — Given PO
Biological: Rituximab — Given IV
Drug: Doxorubicin — Given IV
  Arms: Arm II (frontline chemotherapy, inotuzumab ozogamicin)
Drug: Thioguanine — Given PO
Biological: Inotuzumab Ozogamicin — Given IV
  Arms: Arm II (frontline chemotherapy, inotuzumab ozogamicin)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This partially randomized phase III trial studies the side effects of inotuzumab ozogamicin and how well it works when given with frontline chemotherapy in treating patients with newly diagnosed B acute lymphoblastic leukemia. Monoclonal antibodies, such as inotuzumab ozogamicin, may block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving inotuzumab ozogamicin with chemotherapy may work better in treating young adults with B acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm tolerability of the combination regimen with the addition of inotuzumab ozogamicin to the pediatric-inspired regimen of cancer and leukemia group B (CALGB) 10403.

II. To determine whether the addition of inotuzumab ozogamicin significantly improves the event-free survival (EFS) in patients who achieve an induction response achieved with the pediatric-inspired regimen of CALGB 10403, without censoring for transplant. (Phase III)

SECONDARY OBJECTIVES:

I. To determine the impact of inotuzumab ozogamicin on disease-free (DFS) and overall survival (OS) in patients who achieve an induction response.

II. To determine whether the addition of inotuzumab ozogamicin significantly improves the event-free survival (EFS) in patients who achieve an induction response achieved with the pediatric-inspired regimen of CALGB 10403, with censoring for transplant.

III. To determine the impact of inotuzumab ozogamicin on minimal residual disease (MRD) and correlate this with the EFS, DFS and OS.

IV. To determine the prognosis based on patients' low-density array (LDA) gene signature in terms of EFS, DFS, and OS after treatment with or without inotuzumab ozogamicin when added to the C10403 backbone regimen.

V. To evaluate the toxicity and tolerability of the addition of inotuzumab ozogamicin to the pediatric-inspired regimen of CALGB 10403.

TERTIARY OBJECTIVES:

I. To assess both the correlation of MRD post-induction and at sequential timepoints with LDA signature.

II. To evaluate the influence of MRD status (detectable vs. not and as a continuous measure) in relation to EFS both in the univariate setting as well as adjusting for other clinical features including initial white blood cell (WBC), ethnicity, gender and age at diagnosis.

III. To evaluate the impact of inotuzumab ozogamicin (inotuzumab) on the kinetics of MRD during treatment with inotuzumab in patients randomized to the experimental treatment arm.

IV. To perform genomic analyses to identify and evaluate the incidence and clinical significance of recurring novel fusion genes including those associated with the BCR-ABL1-like signature and to correlate with MRD status, CR rate, EFS and OS.

V. To assess whether rs4958351 is correlated with L-asp allergic reaction in the adolescent and young adult (AYA) population.

VI. To assess the incidence of inherited genetic variants in the GR1A1, CEP72, CPA2, TPMT, NUDT15, GRIN3A, GRIK1, and other genes (which can be found using a whole genome association study [GWAS]), are correlated with increased rates of target toxicities including peripheral neuropathy, hepatotoxicity, pancreatitis, myelosuppression, neurotoxicity, thrombosis, and osteonecrosis, and correlate with treatment discontinuation and other clinical response parameters including complete response (CR) rate, EFS, and OS.

VII. To evaluate asparaginase pharmacokinetics in adolescents and young adults, and investigate its correlation with toxicities and treatment outcomes.

VIII. To investigate the effect of anti-polyethylene glycol (PEG) and anti-agouti signaling protein (ASP) antibodies (PEG-ASP) on ASP enzyme activity.

IX. To measure adherence to oral 6 mercaptopurine (MP) and methotrexate in AYAs with acute lymphoblastic leukemia (ALL) and to examine sociodemographic and behavioral determinants of adherence.

X. To determine the impact of adherence on risk of relapse among AYAs with ALL.

OUTLINE:

COURSE I (REMISSION INDUCTION THERAPY): All patients receive allopurinol orally (PO) once daily until peripheral blasts and extramedullary disease are reduced and cytarabine intrathecally (IT) over 1 minute on day 1. Patients also receive daunorubicin hydrochloride intravenously (IV) and vincristine sulfate IV on days 1, 8, 15 and 22, dexamethasone PO or IV twice daily (BID) on days 1-7 and 15-21, pegylated L-aspiraginase IV on day 4, 5, or 6, and methotrexate IT over 1 minute on days 8 and 29. Patients with central nervous system (CNS) 3 disease receive methotrexate IT over 1 minute also on days 15 and 22. All patients then undergo bone marrow aspirate and biopsy on day 29.

Patients with response to remission induction therapy are randomized to 1 of 2 arms. Patients with no response are omitted from the study.

ARM I:

COURSE II (REMISSION CONSOLIDATION CHEMOTHERAPY): Patients receive cyclophosphamide IV on days 1 and 29, cytarabine IV or SC on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14 and 29-42, and vincristine sulfate IV on days 15, 22, 43, and 50. Patients also receive pegylated L-aspiraginase IV on days 15 and 43, and methotrexate IT on days 1, 8, 15, and 22. Patients with CNS3 receive methotrexate IT only on days 1 and 8. CD20 positive (+) patients receive rituximab IV on days 1, 8, 29, and 36. Patients then undergo bone marrow aspirate and biopsy on day 56.

COURSE III (INTERIM MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 11, 21, 31, and 41, methotrexate IV and IT on days 1, 11, 21, 31, and 41, and pegylated L-aspiraginase IV on days 2 and 22. CD20+ patients receive rituximab IV on days 1 and 11.

COURSE IV (DELAYED INTENSIFICATION): Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50, dexamethasone PO or IV BID on days 1-7 and 15-21, doxorubicin IV on days 1, 8, and 15, and pegylated L-aspiraginase IV on day 4, 5, or 6 and day 43. Patients also receive cyclophosphamide IV on day 29, cytarabine IV or SC on days 29-32 and 36-39, thioguanine PO on days 29-42 and methotrexate IT on days 1, 29, and 36. CD20+ patients receive rituximab IV on days 1 and 8. Patients then undergo bone marrow aspirate and biopsy on day 50.

COURSE V (MAINTENANCE THERAPY): Patients receive vincristine sulfate IV on days 1, 29, and 57, dexamethasone PO or IV BID on days 1-5, 29-33, and 57-61, and mercaptopurine PO on days 1-84. Patients also receive methotrexate IT or PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 12 weeks for up to 3 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive inotuzumab ozogamicin IV on days 1, 8, and 15 and undergo bone marrow aspirate and biopsy on day 28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive remission consolidated chemotherapy, interim maintenance chemotherapy, delayed intensification, and maintenance therapy as in Arm I.

After completion of study treatment, patients are followed up every month for the first year, every 2 months for the second year, every 3 months for the third year, and every 6 months for the fourth through tenth year.

ELIGIBILITY:
Inclusion Criteria:

REGISTRATION ELIGIBILITY CRITERIA (STEP 1)

* Newly diagnosed patients with CD-22 positive B-cell acute lymphoblastic leukemia (WHO criteria) are eligible. Patients with Burkitt type ALL are NOT eligible
* Patients who have BCR-ABL fusion transcript determined by fluorescence in situ hybridization (FISH) or real time-polymerase chain reaction (RT-PCR) or t(9;22)(q34;q11) by cytogenetics are not eligible and should be considered for enrollment on studies that incorporate imatinib during induction; please note: flow cytometry is to be performed at the local reference lab and must include assessment of CD20 and CD22 positivity, as well as CD29 and CD22 anti-positivity
* No prior therapy except for limited treatment (< 7 days) with corticosteroids or hydroxyurea and a single dose of intrathecal cytarabine
* No prior therapy for acute leukemia except emergency therapy (corticosteroids or hydroxyurea) for blast cell crisis, superior vena cava syndrome, or renal failure due to leukemic infiltration of the kidneys; when indicated, leukapheresis or exchange transfusion is recommended to reduce the WBC
* Single-dose intrathecal cytarabine is allowed prior to registration or prior to initiation of systematic therapy for patient convenience; systemic chemotherapy must begin within 72 hours of this intrathecal therapy
* Patients receiving prior steroid therapy are eligible for study; the dose and duration of previous steroid therapy should be carefully documented on case report forms
* Not pregnant and not nursing; for women of childbearing potential only, a negative urine or serum pregnancy test done =< 7 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients with down syndrome are excluded from this study
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN), unless suspected leukemic involvement of the liver
* Direct bilirubin =< 3 x upper limit of normal (ULN), unless suspected leukemic involvement of the liver
* Calculated (calc.) creatinine clearance >= 50 mL/min by Cockcroft-Gault

RANDOMIZATION ELIGIBILITY CRITERIA (STEP 2)

* Completion of remission induction therapy
* Patients with M2 marrow or better are eligible; patients with M3 or M4 marrow (greater than 25% lymphoblasts) will not be eligible to be randomized

  * Rating: M0, M1; Blast Cells (%): 0-5.0
  * Rating: M2; Blast Cells (%): 5.1-25.0
  * Rating: M3; Blast Cells (%): > 25-50
  * Rating: M4; Blast Cells (%): > 50.0
  * The term "blast cell" includes any cell that cannot be classified as a more mature normal element, and includes "leukemic cells," pathologic lymphocytes, and stem cells
* No ascites, effusions or significant edema
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN), except for patients with known Gilbert's syndrome
* Aspartate aminotransferase (AST) =< 8 x upper limit of normal (ULN)
* Completion of first 12 weeks (12+ weeks) of maintenance therapy (Course V)
* Patient has at least 24 weeks (24+ weeks) remaining before end of maintenance therapy (Course V)
* Patient is in complete continuous first remission at entry into A041501-HO1
* Patient is receiving oral anti-metabolite chemotherapy during the maintenance phase of therapy; treatment plan must call for the following doses of antimetabolites: 6MP 75 mg/m2/day orally; methotrexate (MTX) 20 mg/m2/week orally (modification of 6 MP or MTX dosing based on laboratory or clinical parameters is acceptable)
* Patient is able and willing to use the Medication Event Monitoring System (MEMS) TrackCap (e.g. not using a pillbox)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
EFS | Time from induction response to the time of progressive-disease, secondary malignancy, or death, assessed up to 3 years
  Will be compared using log-rank tests. EFS curves will be constructed using the Kaplan-Meier product limit method, and additional analyses will be done using the Cox proportional hazards model. The corresponding hazard ratio, 2- and 3-year EFS estimates will be assessed, and EFS medians along with their 95% confidence intervals for the two treatment arms.

SECONDARY OUTCOMES:
DFS | Time from achievement of CR to the time of relapse and/or death, assessed up to 10 years
OS | Time from randomization to the time of death due to any cause, assessed up to 10 years
  Will be evaluated using Kaplan-Meier as well as Cox regression models.
Proportion of patients who achieve CR or any response to induction therapy | Up to 10 years
  Will be summarized as the proportion of patients who achieve any type of response to induction therapy divided by the number of all evaluable patients registered to this trial and who received at least one dose of induction therapy. Corresponding 95% binomial confidence intervals will also be calculated.
Overall induction response rates | Up to 10 years
  Will be summarized as the proportion of patients who achieve any type of response to induction therapy divided by the number of all evaluable patients registered to this trial and who received at least one dose of induction therapy. Corresponding 95% binomial confidence intervals will also be calculated.
Incidence of adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 | Up to 10 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. In addition, all adverse event data that is graded as 3, 4, or 5 will be reviewed and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The incidence of severe (grade 3+) adverse events or toxicities will be described for each treatment arm, but will also be compared between the arms. Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest between the treatment arms and we will graphically assess differences in maximum grades observed for toxicities between the arms. Tolerability of the treatment arms will be assessed through assessing the number of patients who required dose modifications and/or dose delays.
Proportion of patients who go off treatment due to adverse reactions | Up to 10 years
  Will be assessed within each of the treatment arms and differences explores in these measures between the arms.
Proportion of patients who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial | Up to 10 years
  Will be assessed within each of the treatment arms and differences explores in these measures between the arms.

CONTACTS AND LOCATIONS:
Overall Officials: daniel_deangelo@dfci.harvard.edu J. DeAngelo, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (459):
- United States (454):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Rush MD Anderson Cancer Center at Rush Lisle, Lisle, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Seftel MD. Hyper-CVAD: a regimen for all seasons. Lancet Haematol. 2020 Jul;7(7):e501-e502. doi: 10.1016/S2352-3026(20)30179-4. No abstract available. PMID 32589970